CLINICAL TRIAL: NCT01544946
Title: A Randomized Double-blind Trial Comparing the Effect on Pain of an Oral Sucrose Solution Versus Placebo in Children 1 to 3 Months Old Needing Nasopharyngeal Aspiration
Brief Title: Trial of an Oral Sucrose Solution Versus Placebo in Children 1 to 3 Months Old Needing Nasopharyngeal Aspiration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Serge Gouin, Associate Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sucrose3415
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: pediatrics; emergency medicine; pain; nasopharyngeal aspiration
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sucrose po (Experimental)
  Interventions: Drug: 88% sucrose po
- placebo po (Placebo Comparator)
  Interventions: Drug: placebo po

INTERVENTIONS:
Drug: 88% sucrose po — 88% sucrose solution (Syrup B.P.)
  Arms: sucrose po
Drug: placebo po — sterile water
  Arms: placebo po

SUMMARY:
Background: Early recognition and treatment of pain among children is important for their cognitive development and their future response to pain throughout their life. Oral sweet solutions have been accepted as effective pain reducing agents for procedures in the neonatal population. To date, there have been a limited number of published clinical trials in an emergency setting studying this type of intervention among infants undergoing venous puncture and bladder catheterization. These studies have reported conflicting results. No previous studies have evaluated the utilization of sucrose to manage pain during nasopharyngeal aspiration.

Objective: To compare the efficacy of an oral sucrose solution versus placebo in reducing pain in children one to three months of age during nasopharyngeal aspiration in the Emergency Department.

DETAILED DESCRIPTION:
INTRODUCTION AND JUSTIFICATION

Acute pain is one of the most common adverse stimuli experienced by children, occurring as a result of injury, illness, and necessary medical procedures1. The American Academy of Pediatrics (AAP) and the American Pain Society (APS) have jointly issued a statement promoting the responsibility of paediatricians as leaders and advocates to ensure the humane and competent treatment of pain and suffering in all infants, children, and adolescents.

Long-term effects of unmanaged pain in human infants have been shown to include permanent impairment of elements of cognitive development, such as learning, memory, and behavior, and increased somatisation in childhood. The plasticity of the developing brain and the changes that occur in response to painful stimuli also contribute to altered perceptions of pain later in life. Early painful experiences affect children's future responses to analgesia. Weisman et al found that inadequate analgesia in young children during procedures diminished the effects of adequate analgesia during subsequent procedures. Many studies have suggested that the prompt and accurate recognition and treatment of pain in young infants is important for their immediate comfort and for their best possible lifelong development. Despite the recent interest in paediatric pain assessment, prevention and treatment, many children do not receive adequate management to alleviate pain. The ideal pre-procedural analgesic agent for minor invasive procedures would be a cost-effective, inexpensive, short-acting agent with few associated risks.

The use of sucrose has been well studied for certain procedures in the patients of the neonatal intensive care unit and in the newborn nursery settings, particularly for venous blood draws, capillary blood tests and circumcision. In these studies, infants receiving oral sucrose solutions before procedures cried less and had overall decreased behavioral pain responses when compared with those receiving placebo. Furthermore, sucrose has been shown to be a safe intervention with no serious life-threatening adverse events and only few reported side effects consisting of minimal coughing with administration. Sucrose is inexpensive, short acting, non-sedating, easily administered and non-invasive. Administration of sucrose does not require additional training and does not expose the infant to risks greater than those associated with breast or bottle feeding.

Nasopharyngeal aspiration (NPA) is a common procedure in the Emergency Department (ED), especially during wintertime. It is also a recognized way to support small children with bronchiolitis or upper respiratory viral illness. There is currently a paucity of literature about the perception of pain or discomfort during nasopharyngeal aspiration. Macfarlane and al. compared nasal swab versus nasopharyngeal aspirate for RSV testing in children of 1 month to 20 months. Infant distress was measured using a facial, cry, and movement scoring scale (FLACC). A median score of six was obtaining in the group of nasopharyngeal aspirate in comparison of median score of cinq for nasal swab (p<0,0001).

Sucrose administered by non-nutritive sucking two minutes prior to the procedure is now recognized as a safe16 and efficient way to relieve pain for minor procedures in the neonatal intensive care unit (NICU). It can contribute to decrease the physiologic response to a painful stimulus (heart rate, respiratory rate and decrease in oxygensaturation) as well as attenuate pain behaviors and decrease the overall score in pain scales. Since 1998, the Cochrane Database Review recommends the use of sucrose for procedural pain in the neonatal population. The latest edition (2010) provides sufficient evidence to recommend the use of sucrose for single heel lance punctures and its consideration for venipuncture. Authors conclude that further studies are needed to extend the use of sucrose to some other neonatal common but painful procedures such as bladder catheterization, nasogastric tube insertion and suctioning.

Studies about the use of sucrose for relieving pain in routine immunizations suggest that analgesic properties can have an effect beyond infancy, despite upper age of this limit and appropriate concentration or quantity of sucrose are unknown for this age group. Randomized controlled trials in EDs introduced the use of sucrose for venipuncture or bladder catheterization for older infants. Curtis and al demonstrated a trend toward reducing pain in children of zero to six months of age using sucrose during venipuncture. However the benefit seemed to be limited to infants less than three months old with no significant variation in pain scale scores beyond this age (three to six months). In a second study, Rogers and al. showed that using sucrose while an infant undergoes bladder catheterization reduced variations in pain scale scores and enhanced a quicker return to baseline for infants of 1 to 30 days of life, while infants in the group of 30 to 90 days failed to demonstrate this relation. No specific study was found about pain management during nasopharyngeal aspiration in infants in ED.

Also, studies have used varieties of concentrations of sucrose ranging from 24% to 75%. Systematic reviews of the current literature have been unable to demonstrate superiority of one concentration of a sweet solution over another21-25, but many studies suggested that higher concentrations of sweet solutions seemed more effective. Therefore, the investigators chose to study the effect of a sweet solution named syrup B.P. (product by Laboratoire Atlas inc.) which contains 88% of sucrose. This solution is already commonly used in the population of infants up to three months of age and it is safe (e.g. prednisone syrup or codeine syrup are made using this syrup). A two milliliters dose of 88% sucrose contains the same amount of carbohydrates as 25 milliliters of infant milk formulas which contain approximately 7,5g/100 milliliters 30. Also, 88% sucrose has the same sugar concentration as many other medications which are commonly used in infants, such as oral antibiotics, oral steroid solutions and other pain medications (e.g. codeine syrup). This syrup is of particular interest as it is of low cost ($9,58 for a bottle of 2000 milliliters), universally available, stable and viable for approximately three months. Therefore, the procedure studied here would be easy to apply in most clinical settings.

Finally, the painful procedure chosen for the study is nasopharyngeal aspiration. This procedure is frequently performed in the ED in this age group, particularly in the winter either as a therapeutic or diagnostic procedure.

To date, there are no pain scales which have been validated precisely for the age group studied in this project. However, the Face, Legs, Activity, Cry and Consolability (FLACC) scale is recommended by the IMMPACT group (Initiative on Methods, Measurement and Pain Assessment in Clinical Trials). FLACC is an easily applicable pain scale in which the observer scores a patient on five categories, from zero to two points, for a total score of maximum 10 points. The validity and reliability of this pain scale has been established in the past for children from 2 months to 7 years. Validity was evaluated by comparing the FLACC scale with the Objective Pain Scale and demonstrated that both tools showed similar behaviours (r=0.80; p<0.001). The interrater reliability between two observers was considered good (r[87]=0.94; p<0.001) with a kappa value greater than 0,50 for each category. Therefore, this pain scale was chosen as the measure of the investigators primary outcome, in this population of infants from one to three months old. Furthermore, the Neonatal Infant Pain Scale (NIPS)is a well validated pain scale for newborns up to one month of age. This pain scale was chosen as a secondary outcome. The investigators hypothesize that using one pain scale validated in infants up to 1 month of age and another validated in infants older than two months of age will allow us to assess pain in infants from one to three months of age best, given current available tools. Furthermore, several other patient parameters will be used to corroborate findings.

HYPOTHESIS

The investigators believe that providing an oral sucrose solution during nasopharyngeal aspiration will decrease pain levels in infants one to three months of age.

OBJECTIVES

The investigators primary objective is to compare the efficacy an oral 88% sucrose solution to a placebo solution in reducing pain as assessed by the FLACC scale in children of one to three months during nasopharyngeal aspiration in the ED. The investigators secondary objectives are to asses changes in pain levels as per the NIPS scores. The investigators will also measure variations of heart rate and crying time. Any side effects will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Infants from one to three months (one month or more but less than three months old) of actual age (not corrected) requiring a nasopharyngeal aspiration as a part of their planned ED management during weekdays from 8h to 16h.

Exclusion Criteria:

* Preterm infants (i.e. born <37 weeks)
* Chronic cardio-pulmonary condition
* Assisted ventilation (such as tracheostomy or oxygen dependance)
* Technology dependant (such as enteral feeding tubes)
* Oropharyngeal malformation or dysfunction (such as cleft palate or micrognatia)
* Previous participation in this study
* Painful procedures in the preceding 60 minutes (bladder catheterization, vesical puncture, lumbar puncture, capillary blood tests)
* Parental language barrier (French and/or English)

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Difference in pains scores related to nasopharyngeal aspiration | one minute

SECONDARY OUTCOMES:
Difference in pain scores related to nasopharyngeal aspiration | 3 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gouin, MDCM, FRCPC, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada